CLINICAL TRIAL: NCT07089056
Title: Effects of Transcranial Direct Current Stimulation After Short-term Immobilization on Motor Learning and Hand Function in Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023145H
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Transcranial Direct Current Stimulation
Keywords: Transcranial direct current stimulation; immobilization; motor learning
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Immobilization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immobilization and Transcranial Direct Current Stimulation (Experimental): The participants' right hands will be immobilized for 16 hours, and they will receive 20 minutes of transcranial direct current stimulation before the immobilization period ends.
  Interventions: Device: sham transcranial direct current stimulation; Procedure: immobilization
- Immobilization and Sham Transcranial Direct Current Stimulation (Experimental): The participants' right hands will be immobilized for 16 hours, and they will receive 20 minutes of transcranial direct current stimulation before the immobilization period ends.
  Interventions: Procedure: transcranial direct current stimulation; Procedure: immobilization
- Blank control group (No Intervention)

INTERVENTIONS:
Procedure: transcranial direct current stimulation — The intervention will be conducted using a battery-powered stimulator (TCS-E2000, Shenzhen Yingchi Technology Co., Ltd) through a pair of saline-soaked sponge electrodes (5 cm × 5 cm).The stimulation intensity will be set at 2 mA. The stimulation will last for 20 minutes, with a 10 s fade-in period at the start and a 10-s fade-out period at the end of stimulation. The anodal electrode will be placed over the primary motor cortex (M1), and the reference electrode will be positioned at the center of the forehead.
  Arms: Immobilization and Sham Transcranial Direct Current Stimulation
Device: sham transcranial direct current stimulation — The intervention will be conducted using a battery-powered stimulator (TCS-E2000, Shenzhen Yingchi Technology Co., Ltd) through a pair of saline-soaked sponge electrodes (5 cm × 5 cm).The stimulation intensity will be set at 2 mA. The anodal electrode will be placed over the primary motor cortex (M1), and the reference electrode will be positioned at the center of the forehead for 20 minutes. However, there will be current only during the first 10 seconds and the last 10 seconds.
  Arms: Immobilization and Transcranial Direct Current Stimulation
Procedure: immobilization — The researchers will use an upper limb fixation splint to fix the right upper limb of the participants, with the elbow joint flexed at 90 degrees, to ensure that all movements of the wrist, metacarpophalangeal joints, proximal interphalangeal joints, and interphalangeal joints are completely restricted. To avoid discomfort caused by the splint, soft bandages will be wrapped around the hand, and the splint will be adjusted to fit the shape of the hand. Ensure that the fingertips are visible to ensure good blood circulation. The subjects need to wear the upper limb fixation splint for 16 hours. Instruct the subjects to minimize movement and use of the right upper limb as much as possible. During the immobilization process, pay attention to checking if the participants have numbness or other discomfort, as well as whether the blood flow is good. If any adverse symptoms occur, the immobilization will be immediately terminated.
  Arms: Immobilization and Sham Transcranial Direct Current Stimulation; Immobilization and Transcranial Direct Current Stimulation

SUMMARY:
The purpose of the study is to investigate the effects of short-term braking on the motor learning and fine motor skills of healthy adults, and to analyze whether transcranial direct current stimulation can alleviate the effects of braking on motor learning and fine motor skills.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effects of 16-hour short-term immobilization on the motor learning and fine motor skills of healthy adults, and to analyze whether transcranial direct current stimulation intervention can alleviate the effects of immobilization on motor learning and fine motor skills.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 18 and 25 years;
* (2) normal or corrected-to-normal vision;
* (3) right-handedness.

Exclusion Criteria:

* (1) with history of pregnancy, cardiovascular disease, other physical impairments or illnesses;
* (2) with personal or family history of mental illness;
* (3) implanting any internal or external medical devices;

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-21 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Sequence Reaction Time Task | Baseline; after one week
  The participants will sit in front of the laptop and placed their four right fingers on the four keys on the keyboard. In this task, a white circle appears above one of four horizontally arranged white squares on the computer screen with black background. Participans will be instructed to press the proper button on the response pad (buttons H, J, K, L) using the corresponding finger of the right hand (index finger for button H, middle finger for button J, ring finger for button K, and small finger for button L) when the white circle appeared at the left side, middle-left side, middle-right side, or right side of the computer screen, respectively. Each session consists of eight blocks, with each block comprising 120 trials.

SECONDARY OUTCOMES:
Purdue Pegboard Test | Baseline; after one week
  The Purdue Pegboard (model 32020; Lafayette Instrument Co., Lafayette,Indiana) performed the tests. The nail jacks were arranged in two parallel columns, and the nail, washer, and collar were placed in the four cups at the top of the plate before the experiment began. Subjects will be prompted to begin the test by using a nail to jack first with their right hand, then with their left hand, and finally with both hands simultaneously. Each segment was 30 s in duration, and the number of nails transferred by the participant was recorded. Finally, participants will assemble a nail, a washer, a collar and a washer on top of it, starting with their right hand in 1 minute. Each of the above sections was repeated three times to obtain an average score.
Reach and grasp action test | Baseline; after one week
  The reach and grasp test included two parts: the fine grasp test and the gross grasp test. In the fine grip test, participants will be instructed to grasp a pencil with the tips of their thumb and index finger, and in the coarse grip test, they are instructed to grasp a tennis ball with their entire hand. Participants will seat in front of a table, and the tester placed the objects on the marked points. Participants began and ended the grasp task at the same location (30cm from the marker), and all performed the same posture (index finger in contact with thumb). Participants will complete the grasp task 15 times at their own pace.
  Infrared motion capture system will be used to record 3D kinematic data during the reaching and grasping movements.